CLINICAL TRIAL: NCT00618800
Title: Preventing Falls Through Enhanced Pharmaceutical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Susan Blalock, PhD, Associate Profesor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5-38047/0-401-4974
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Falls
Keywords: Falls; Elderly; Injury; Medication; Pharmacy; Pharmacist
MeSH Terms: conditions — Wounds and Injuries | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist Care (Experimental): Pharmacist Intervention
  Interventions: Behavioral: Pharmaceutical Care
- Control (Active Comparator): Written information only group
  Interventions: Other: Written Materials

INTERVENTIONS:
Behavioral: Pharmaceutical Care — Participants receive written information about falls prevention and a personal consultation from a community pharmacist concerning their medication regimen. The pharmacist follows up, as required, with participants' physicians to coordinate any recommended medication changes.
  Arms: Pharmacist Care
Other: Written Materials — Participants receive written information about falls prevention.
  Arms: Control

SUMMARY:
The objective of the proposed study is to reduce the incidence of falls and fall-related injuries among community-dwelling older adults by better utilizing community pharmacists to advise patients and physicians on medication management.

DETAILED DESCRIPTION:
Falls are the leading cause of both fatal and nonfatal injuries among older adults in the United States. Past research suggests that individuals taking four or more prescription medications are at increased risk for falls. CNS-active drugs (e.g., benzodiazepines), in particular, have been associated with increased risk. Research also suggests that interventions to reduce inappropriate medications can reduce the risk of falls. This finding comes primarily from multifaceted interventions, however, and the impact of medication modification, by itself, remains largely unknown.

This study is using a a randomized controlled clinical trial design to evaluate a falls prevention program targeting community-dwelling older adults through community pharmacies. The study focuses on individuals at high risk for future falls. Individuals in the intervention group receive an in-depth consultation concerning their current medications, conducted by a community pharmacist. The consultation is designed to elicit medication-related problems (e.g., orthostatic hypotension, daytime sedation). Problems identified during the consultation, and therapeutic recommendations designed to address these problems, are communicated to the prescribing physician. With physician approval, appropriate modifications are made to the patient's medication regimen. The primary study endpoints are: time to first fall and proportion of individuals who fall during the one-year follow-up period.

Two primary hypotheses will be tested.

1. Compared to individuals in the control group, individuals in the intervention group will experience a 30% reduction in the hazard of falling (hazard ratio=0.70) for time to first fall following randomization.
2. Compared to individuals in the control group, 25% fewer people in the intervention group will experience a fall during the one-year follow-up period.

If the intervention is effective in reducing falls, these effects should be mediated by improvements in the overall quality of medication use. Thus, we will also assess effects of the intervention on: change in the number of inappropriate medications prescribed and change in the number of CNS-active medications prescribed.

One secondary hypotheses will be tested.

1. Compared to individuals in the control group, individuals in the intervention group will experience a 40% reduction in the use of high-risk medications during the one-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Currently taking at least four prescription medications
* Currently taking at least one high risk medication
* At least one fall during 12 month period before study entry
* Able to speak and read English

Exclusion Criteria:

* Resident of a long-term care facility
* Cognitive impairment
* Housebound

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-08; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time to first fall | One Year
Proportion of participants who fall | One Year

SECONDARY OUTCOMES:
Use of high-risk medications | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Blalock, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Injury Prevention Research Center, Chapel Hill, North Carolina, United States